CLINICAL TRIAL: NCT01108666
Title: Phase I Dose Escalation Trial of Proton Beam Radiotherapy With Concurrent Chemotherapy and Nelfinavir for Inoperable Stage III NSCLC
Brief Title: Proton Beam Radiation With Concurrent Chemotherapy and Nelfinavir for Inoperable Stage III Non Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01510
Record Dates: First submitted 2010-04-12; First posted 2010-04-22 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Stage IIIA or IIIB NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton RT and Nelfinavir (Experimental)
  Interventions: Drug: Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir — Two dose levels of Nelfinavir will be evaluated in each concurrent chemotherapy group (carboplatin/paclitaxel and cisplatin/etoposide) at the RPTD does of proton beam radiotherapy: 625 and 1250 mg PO bid.

SUMMARY:
Seventy two patients are being asked to take part in this research study because they have been diagnosed with Stage IIIA or IIIB non-small cell lung cancer (NSCLC). This study is being done to determine the highest safe dose of proton beam radiotherapy and/or study drug (called Nelfinavir) that can be given with concurrent chemoradiotherapy to patients with cancer without causing bad side effects; and to develop biomarker for clinical outcome. This study will be done in two phases. In the first phase, feasibility will be established. We will follow patients treatment courses and record side effects at the standard proton radiation dose that can be given together with Cisplatinum + Etoposide or Carboplatin + Paclitaxel. In the second phase, we will see if it is possible to increase the total proton radiation dose or study drug without increasing the number of bad side effects while treated together with chemotherapy drugs.

DETAILED DESCRIPTION:
Overall objectives:

1. Determine MTD of proton beam radiotherapy with concurrent cisplatin and etoposide for stage III NSCLC.
2. Determine MTD of proton beam radiotherapy with concurrent carboplatin and paclitaxel for stage III NSCLC in non-cisplatin candidates.
3. Determine MTD of Nelfinavir with concurrent chemoradiotherapy for stage III NSCLC at RPTD of proton beam radiotherapy.
4. Develop biomarker for clinical outcome with concurrent chemoradiotherapy in stage III NSCLC.
5. To determine clinical efficacy, as defined by metabolic response, sites of recurrence (e.g., local, regional, distant) and progression-free and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of NSCLC.
2. Stage IIIA or IIIB NSCLC.
3. Patients must have no evidence of metastatic disease based on routine imaging.
4. Patients must have a Karnofsky Performance Status of 60.
5. Age 18 and older.
6. Patients must be able to provide informed consent.
7. Adequate bone marrow function (i.e. WBC larger than or equal to 4000/mm3, platelets larger than or equal to 100,000 mm3).
8. Adequate renal function for cisplatin or carboplatin as determined by the medical oncologist: Usually Calculated creatinine clearance (CrCl) larger than or equal to 45 mL/min or serum creatinine level smaller than or equal to1.5 x institutional ULN.
9. Patients must have bilirubin 1.5 mg/dl.
10. Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms or other barrier methods etc).
11. Hysterectomy or menopause must be clinically documented.

Exclusion Criteria:

1. Prior or simultaneous malignancies within the past two years (other than cutaneous squamous or basal cell carcinoma or melanoma in situ).
2. Pregnant women, women planning to become pregnant and women that are nursing.
3. Actively being treated on any other research study.
4. For the Nelfinavir phase of the trial only: Patients who are taking Antiarrhythmics (amiodarone, quinidine), Antimycobacterial (rifampin), Ergot Derivatives (dihydroergotamine, ergonovine, ergotamine, ethylergonovine), Herbal Products (St. John's wort/ hypericum perforatum), HMG-CoA Reductase Inhibitors (lovastatin, simvastatin), Neuroleptic (pimozide), Proton Pump Inhibitors, or Sedative/ Hypnotics (midazolam, triazolam). Note: Patients with the following conditions are deemed unsuitable for cisplatin-based chemotherapy (and will be treated with carboplatin): (a) Hearing impairment/ peripheral neuropathy Grade 1 or less at baseline (b) Symptomatic/uncontrolled congestive heart failure (unable to tolerate volume load with pre- and post-cisplatin hydration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-03; Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton RT and Nelfinavir
Started | 7 (Despite all possible efforts to contact the PI/study, data per dose-level are not available to be reported)
Completed | 7 (Despite all possible efforts to contact the PI/study, data per dose-level are not available to be reported)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Despite all possible efforts to contact the PI/study, data per dose-level are not available to be reported
Arm/Group | Proton RT and Nelfinavir
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.11 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Proton Radiation
Description: Ability to successfully plan proton plans
Time Frame: 10 days
Population: The PI has left the institution and despite all possible efforts is not able to be contacted, data are not available to be reported.
Arm/Group | Proton RT and Nelfinavir
Number analyzed (Participants) | 0

2. Primary Outcome: Acute Toxicity (or Dose Limiting Toxicity)
Description: Dose limiting toxicities of grade 3 or higher per CTCAE 4.0
Time Frame: 14 days
Population: The PI has left the institution and cannot be contacted despite all possible efforts, data are not available to be reported.
Arm/Group | Proton RT and Nelfinavir
Number analyzed (Participants) | 0

3. Primary Outcome: Late Toxicity
Description: Late toxicities graded according to the RTOG/EORTC late morbidity scale
Time Frame: 5 years
Population: Despite all possible efforts to contact the PI/study team members, no data are available to be reported
Arm/Group | Proton RT and Nelfinavir
Number analyzed (Participants) | 0

4. Secondary Outcome: Clinical Efficacy
Description: Defined as metabolic response (complete, partial or less than partial) based on PET/CT imaging. Patients are followed for disease recurrence and site (local, regional, distant). Progression-free and overall survival are defined as from start of treatment to first documented recurrence (for PFS), date of death or last patient contact alive.
Time Frame: One year
Population: as for outcome 2
Arm/Group | Proton RT and Nelfinavir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 days
Description: Despite all possible efforts to contact the PI/study, data per dose-level are not available to be reported
Arm/Group | Proton RT and Nelfinavir
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton RT and Nelfinavir (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1
Hypotension (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton RT and Nelfinavir (N=7)
Anemia (Blood and lymphatic system disorders) | 5
Hypotension (Cardiac disorders) | 1
Other Ear and labyrinth disorders (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 4
Esophageal pain (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 4
Gastroparesis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral dysesthesia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 5
Fever (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pharyngolaryngeal pain (General disorders) | 1
Alopecia (Immune system disorders) | 1
Esophageal infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Mucosal infection (Infections and infestations) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Reproductive system and breast disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT01108666/Prot_SAP_000.pdf